CLINICAL TRIAL: NCT05704647
Title: Phase II Study of Nivolumab in Combination With Relatlimab in Patients With Active Melanoma Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1203; NCI-2023-00571 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma | interventions — relatlimab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relatlimab+Nivolumab (Experimental): Participants will receive nivolumab in combination with relatlimab by vein over about 30 minutes on Day 1 of each 28-day study cycle. You may receive up to 25 doses of the study drugs.
  Interventions: Drug: BMS-986213 (Relatlimab-Nivolumab FDC); Drug: Nivolumab; Drug: Relatlimab

INTERVENTIONS:
Drug: BMS-986213 (Relatlimab-Nivolumab FDC) — Given by IV (vein)
  Other Names: Relatlimab; BMS-986016
Drug: Nivolumab — Given by IV (vein)
Drug: Relatlimab — Given by IV (vein)

SUMMARY:
To learn if giving nivolumab in combination with relatlimab can help to control melanoma that has spread to the brain (melanoma with brain metastases). The safety and side effects of the study drug combination will also be studied.

DETAILED DESCRIPTION:
Primary Objectives:

• To assess the intracranial objective response rate (iORR), defined as intracranial CR + PR per modified RECIST 1.1 criteria, of nivolumab + relatlimab (nivo+rela) in subjects with MBM and treatment naïve to anti-PD-1 agents in the metastatic setting.

Secondary Objectives:

* To determine the safety of the combination of nivo+rela
* To assess the clinical benefit rate (CBR), defined as CR + PR + SD >6 months, of the combination
* To determine overall response rates (intracranial + extracranial), DoR, PFS, and using a modified version of iRANO and compared to modified RECIST v1.1 and Response Assessment in Neuro-oncology - Brain Metastases (RANO-BM) for patients treated with nivo+rela
* To determine the 1-year intracranial progression-free survival rate for the combination of nivo+rela
* To determine overall survival
* Advanced MRI imaging to assess for edema, tumor response, and predictors of response and radiation necrosis
* To evaluate the brain-specific safety and tolerability of the combination regimen in subjects with or without SRT received prior to study entry, or on study
* To evaluate changes in neurocognitive function and health-related quality of life
* To assess available tumor tissue - intracranial and/or extra cranial - in specimens obtained at baseline (archival and/or fresh tissue), on treatment, and at time of progression
* To assess immune cell subsets by flow cytometry, TCR NGS for diversity and clonality, cytokine expression, cfDNA from peripheral blood.

Exploratory Endpoints:

* Radiotherapy-assisted PFS defined as time from study treatment initiation to the first occurrence of disease progression or death from any cause, whichever occurs first, as determined by the investigator according to RECIST v1.1 modified by excluding ≤ 5 lesions that can be treated by SRT from the sum of largest diameters from baseline onwards.
* To explore the association between baseline and on-treatment gut microbiome features with response and toxicity
* To understand the association between habitual diet and gut microbiome features in this study population.
* To explore predictors of biological response through the change in metabolic parameters

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Life Expectancy > 12 weeks.
3. Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.

   • Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study.
4. Histologically confirmed malignant melanoma with measurable metastases in the brain (≥ 0.5 cm).
5. At least one measurable intracranial target lesion, which previously was not treated with local therapy (no prior SRS to this lesion).

   • Largest diameter of ≥ 0.5cm, but ≤ 3cm as determined by contrast-enhanced MRI.
6. Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (blocks are preferred) OR at least 4 unstained slides, with an associated pathology report, for testing of tumor PD-L1 expression:

   * Tumor tissue should be of good quality based on total and viable tumor content.
   * Patients who do not have tissue specimens may undergo a biopsy during the screening period. Acceptable samples include core-needle biopsies for deep tumor tissue or excisional, incisional, punch, or forceps biopsies for cutaneous, subcutaneous, or mucosal lesions. Fine Needle Aspirations (FNA) will not be considered acceptable for tissue procurement.
   * Tumor tissue from bone metastases is not evaluable for PD-L1 expression and is therefore not acceptable.
   * However, if repeat biopsy is not feasible, and no archival tissue available patient still may be enrolled.
7. Prior SRT and prior excision of up to 5 MBM is permitted if there has been complete recovery, with no neurologic sequelae, and measurable non irradiated lesions remain.
8. Growth or change in a lesion previously irradiated will not be considered measurable. Regrowth in cavity of previously excised lesion will not be considered measurable.

   • Any prior SRT to brain lesions or prior excision must have occurred ≥ 1 weeks before the start of dosing for this study.
9. Radiation to NON-CNS lesions. Prior radiation to NON-CNS is allowed and does not require a washout period for treatment initiation.
10. Subjects must be free of neurologic signs and symptoms related to metastatic brain lesions and must not have required or received systemic corticosteroid therapy in the 5 days prior to beginning protocol therapy.
11. ECOG performance status ≤1.
12. Adequate organ function as described below.
13. Women of child-bearing potential (WOCBP) must not be breastfeeding and must have a negative pregnancy test within 3 days prior to initiation of dosing. She must agree to use an acceptable method of birth control from the time of the negative pregnancy test, through the duration of treatment with the study combination plus 5 half lives of study treatment for a total of 5 months post -treatment completion. WOCBP must agree to adhere to the contraceptive guidance in Appendix 5. NOTE: A female participant is eligible to participate if she is not a woman of childbearing potential as defined Appendix 4.
14. All associated toxicity from previous or concurrent cancer therapy must be resolved (to ≤ grade 1 or baseline) prior to study treatment administration. This excludes non-serious toxicities. However, stable endocrinopathies requiring replacement therapy will be allowed.
15. Steroids for physiological replacement are allowed.

Exclusion Criteria:

1. History of known leptomeningeal involvement (lumbar puncture not required).
2. Previous stereotactic or highly conformal radiotherapy within 1 weeks before the start of dosing for this study. NOTE: The stereotactic radiotherapy field must not have included the brain index lesion(s).
3. Subjects previously treated with SRT > 5 lesions in the brain. Prior whole brain radiation is not allowed.
4. Brain lesion size > 3 cm.
5. Prior checkpoint inhibitor therapy in the metastatic setting

   • Patients who received ipilimumab and/or anti-PD1 as adjuvant or neoadjuvant therapy must have a 6-month washout before receiving any dosing on this study.
6. Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
7. Subjects with major medical, neurologic or psychiatric condition who are judged as unable to fully comply with study therapy or assessments should not be enrolled.
8. Subject has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. Note: The time requirement does not apply to participants who underwent successful treatment of superficial bladder cancer, in situ cervical cancer, or other in-situ cancers. Subjects with a completely treated prior malignancy and no evidence of disease for ≥ 2 years are eligible.

   a. Skin Cancer Exclusion: Please note that basal cell carcinoma and squamous cell carcinoma is exempt from needing resection prior to treatment. (Resection can be completed after the start of treatment).
9. Has a known history of or is positive for hepatitis B (hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (hepatitis C virus [HCV] RNA [qualitative] is detected).

   a. NOTE: Without known history, testing needs to be performed to determine eligibility. Hepatitis C antibody (Ab) testing is allowed for screening purposes in countries where HCV RNA is not part of standard of care.
10. Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.
11. The use of corticosteroids is not allowed for 10 days prior to initiation of therapy (based upon 5 times the expected half-life of dexamethasone) except patients who are taking steroids for physiological replacement. If alternative corticosteroid therapy has been used, consultation with the PI is required to determine the washout period prior to initiating study treatment.
12. Subjects with a condition requiring systemic treatment with either corticosteroids (≤ 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study initiation. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
13. Major surgical procedure, open biopsy (excluding skin cancer resection), or significant traumatic injury within 14 days of initiating study drug (unless the wound has healed) or anticipation of the need for major surgery during the study.
14. Non-healing wound, ulcer, or bone fracture.
15. Women who are breast-feeding or pregnant.
16. Uncontrolled intercurrent illness (i.e., active infection ≥ grade 2) or concurrent condition that, in the opinion of the Investigator, would interfere with the study endpoints or the subject's ability to participate.
17. History of clinically significant cardiac disease or congestive heart failure > New York Heart Association (NYHA) class 2. Subjects must not have unstable angina (anginal symptoms at rest) or new-onset angina within the last 3 months or myocardial infarction within the past 6 months or a history of myocarditis.
18. Troponin T (TnT) or I (TnI) > 2 × institutional ULN. Participants with TnT or TnI levels between > 1 to 2 × ULN will be permitted if repeat levels within 24 hours are ≤ 1 ULN. If TnT or TnI levels are between >1 to 2 × ULN within 24 hours, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2 × ULN, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. Notification of the decision to enroll the participant following cardiologist recommendation has to be made to the principal investigator.
19. Investigational drug use within 14 days (or 5 half-lives, whichever is longer) of the first dose of nivolumab and relatlimab.
20. With a history of non-infectious pneumonitis that required steroids or current pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Tawbi, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org